CLINICAL TRIAL: NCT03862105
Title: Pilot Testing for Post-Cystectomy mHealth Tool to Improve Perioperative Care
Brief Title: Testing the Utilization of a Mobile Health App for Patients Undergoing Cystectomy Surgery for Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC1856
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Invasive Bladder Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health App with Provider Monitoring/Care (Experimental): 30 patients enrolled by the study team will receive notifications through a mobile health app (Twistle) before and after surgery. Patient Reported Outcome data will be collected through patient responses in this app and timely clinician feedback will be provided to patients to prevent complications and readmission.
  Interventions: Other: Mobile Health app tool - Twistle

INTERVENTIONS:
Other: Mobile Health app tool - Twistle — The investigators propose to use radical cystectomy as a model to examine the utilization of an electronic, internet-based mobile health intervention that can prospectively collect Patient Reported Outcome data while providing timely feedback to patients and clinicians. This mobile health intervention will utilize a well-established platform (Twistle) that can be accessed through multiple technologies, including laptops, smartphones, and other computer-based systems.

SUMMARY:
This is a pilot study that involves human subjects undergoing cystectomy surgery for bladder cancer, testing the utilization of a mobile health app that promotes postoperative patient engagement, along with provider monitoring and care. The aim of this pilot study is to assess feasibility and acceptability of an Internet-based mobile health tool following cystectomy discharge. Objectives will be met by assessing weekly adherence, determining acceptability of mobile health questions post-surgery by patients and providers, and by obtaining participant feedback regarding the tool. Complications, re-admissions, and resource utilization will also be monitored throughout the study. The hypothesis is that an mobile health intervention that tracks PROs, provides educational content, and allows real-time feedback via internet-enabled devices has the potential to improve the quality of care delivery and overall patient experience following surgery by decreasing resource utilization and improving symptom control and communication.

DETAILED DESCRIPTION:
Radical cystectomy will be used as a model to examine the utilization of an electronic, internet-based mobile health intervention that can prospectively collect PRO data while providing timely feedback to patients and clinicians. This mobile health intervention will utilize a well-established platform (Twistle) that can be accessed through multiple technologies, including laptops, smartphones, and other computer-based systems. The objective is to evaluate the feasibility of pre-specified Patient Reported Outcomes and educational content in an existing mobile health communications platform which tracks patient symptoms and provides real-time feedback to patients and providers following cystectomy discharge. Patient Reported Outcome questions and responses will be inputted using validated questions with branching logic to drive feedback based upon responses. The intent of this study is to evaluate feasibility and acceptability of this mobile health tool following cystectomy discharge. Usual care will continue in coordination with this intervention.

ELIGIBILITY:
Minimum Age: 18 Years Maximum Age: 99 Years Sex: All Gender Based: No

Criteria: Inclusion Criteria:

* Male or female patients with invasive bladder cancer scheduled for radical cystectomy at UNC within the next 30 days
* English-speaking
* Ability to access the Internet (either themselves or with assistance from their caregiver)
* Ability to read
* Ability to provide informed consent.

Exclusion Criteria:

* Inability to read
* Inability to provide informed consent
* Severe psychiatric illness
* Cystectomy surgery without cancer diagnosis
* Non-English speaking

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of the tool (Twistle): percentage of patients using the tool at least once weekly | 90 days postoperative
  percentage of patients using the tool at least once weekly

SECONDARY OUTCOMES:
Acceptability of tool (Twistle): Percentage of patients being satisfied or very satisfied with the mobile health tool | 90 days postoperative
  Percentage of patients being satisfied or very satisfied with the mobile health tool, determined through an online post-intervention survey, addressing ease of use, convenience, privacy and confidentiality, and willingness to use the tool.

CONTACTS AND LOCATIONS:
Overall Officials: Angela B Smith, MD,MS,FACS, Principal Investigator — Associate Professor, Dept of Urology, Director of Urologic Oncology
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials